CLINICAL TRIAL: NCT04163679
Title: Combining Vaginal Preparation and Azithromycin in Reduction of Post Cesarean Infections: A Randomized Controlled Trial
Brief Title: Vaginal Preparation and Azithromycin to Reduce Post Cesarean Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment issues
Sponsor: Womack Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen L Wilson, Program Director of Obstetrics and Gynecology Residency Chief of Maternal Fetal Medicine and Obstetrics Chief, Womack Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHC-A-19-033
Record Dates: First submitted 2019-11-08; First posted 2019-11-15 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Infection; Obstetric Labor Complications; Endometritis; Cesarean Delivery Affecting Fetus; Wounds Injuries
MeSH Terms: conditions — Infections; Obstetric Labor Complications; Endometritis; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Preparation (Experimental): In addition to standard care, subjects will undergo vaginal preparation (VP). A VP kit includes sponge sticks and sponges soaked in a povidone-iodine 10% solution.
  Interventions: Procedure: Vaginal Preparation
- Standard Infection Procedures (Sham Comparator): The very staff will follow hospital protocols for the cesarean delivery. The subject and the infant will be provided care in accordance with current medical standards and be discharged at the discretion of the attending physician.
  Interventions: Procedure: Vaginal Preparation

INTERVENTIONS:
Procedure: Vaginal Preparation — One sponge stick will be inserted into the vagina, where it will stay during the scrubbing of thighs and genitals.
  One sponge will be used to scrub the right inner thigh from mid-thigh to right labia majora. This sponge will then be discarded.
  A second sponge will be used to scrub the left inner thigh from mid-thigh to left labia majora. This sponge will then be discarded.
  A third sponge will be used to scrub the mons pubs, labia majora and minor, perineum and rectum in that order then will be discarded. This will be repeated with a fourth sponge.
  The existing sponge stick in the vagina will be rotated in the vagina twice then removed. This will be discarded.
  A second sponge stick will be inserted in the vagina, rotated twice then removed. As it is removed from the vagina, the perineum and rectum will be swabbed with the stick in that order then discarded. This will be repeated using a third sponge stick.

SUMMARY:
asdgf

DETAILED DESCRIPTION:
asdf

ELIGIBILITY:
Inclusion Criteria:

* full term pregnancy
* undergoing labored, non-emergent cesarean section
* patient in labor

Exclusion Criteria:

Azithromycin contraindicated:

* Known hypersensitivity to azithromycin, erythromycin, macrolides or ketolide medications.
* liver dysfunction
* Prescription medications which may interact with azithromycin, such as nelfinavir or warfarin
* A history of a cardiac dysrhythmia (irregular heartbeats)
* Known hypersensitivity to iodine
* Patients carrying fetuses with known congenital anomalies
* Immunodeficiency
* Patients who are not in labor at the time of delivery
* Non-english speaking subjects or subjects with language barriers

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females admitted to Womack Army Medical Center who deliver full term via unscheduled, non-emergent cesarean section following labor
Enrollment: 84 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Infection rates | Six weeks postpartum
  wound infection
Infection rates | six weeks postpartum
  endometritis

SECONDARY OUTCOMES:
Infant Birth Weight | Four weeks after birth
  record their birth weight (gm)
Infant Apgar scores | Four weeks after birth
  Apgar scores
Infant Length of hospital stay | Four weeks after birth
  Hospital stay (days)
Numbers of Infants admitted to NICU | four weeks after birth
  Infant admission to neonatal intensive care unit
Number of Infants that develop respiratory distress | Four weeks after birth
  The infant acquiring the condition of respiratory distress
Number of Infants that develop sepsis | Four weeks after birth
  Infant acquiring sepsis
Number of infants that die | Four weeks after birth
  Infant death

CONTACTS AND LOCATIONS:
Locations (1):
- Womack Army Medical Center, Fort Bragg, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mackeen AD, Packard RE, Ota E, Berghella V, Baxter JK. Timing of intravenous prophylactic antibiotics for preventing postpartum infectious morbidity in women undergoing cesarean delivery. Cochrane Database Syst Rev. 2014 Dec 5;2014(12):CD009516. doi: 10.1002/14651858.CD009516.pub2. PMID 25479008
- [Result] Conroy K, Koenig AF, Yu YH, Courtney A, Lee HJ, Norwitz ER. Infectious morbidity after cesarean delivery: 10 strategies to reduce risk. Rev Obstet Gynecol. 2012;5(2):69-77. PMID 22866185
- [Result] Tita AT, Szychowski JM, Boggess K, Saade G, Longo S, Clark E, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Abramovici A, Ambalavanan N, Cutter G, Andrews W; C/SOAP Trial Consortium. Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. N Engl J Med. 2016 Sep 29;375(13):1231-41. doi: 10.1056/NEJMoa1602044. PMID 27682034
- [Result] Tuuli MG, Liu L, Longman RE, Odibo AO, Macones GA, Cahill AG. Infectious morbidity is higher after second-stage compared with first-stage cesareans. Am J Obstet Gynecol. 2014 Oct;211(4):410.e1-6. doi: 10.1016/j.ajog.2014.03.040. Epub 2014 Mar 18. PMID 24657794
- [Result] Kawakita T, Landy HJ. Surgical site infections after cesarean delivery: epidemiology, prevention and treatment. Matern Health Neonatol Perinatol. 2017 Jul 5;3:12. doi: 10.1186/s40748-017-0051-3. eCollection 2017. PMID 28690864
- [Result] Tita AT, Hauth JC, Grimes A, Owen J, Stamm AM, Andrews WW. Decreasing incidence of postcesarean endometritis with extended-spectrum antibiotic prophylaxis. Obstet Gynecol. 2008 Jan;111(1):51-6. doi: 10.1097/01.AOG.0000295868.43851.39. PMID 18165392
- [Result] Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. Cochrane Database Syst Rev. 2014 Oct 28;2014(10):CD007482. doi: 10.1002/14651858.CD007482.pub3. PMID 25350672
- [Result] Caissutti C, Saccone G, Zullo F, Quist-Nelson J, Felder L, Ciardulli A, Berghella V. Vaginal Cleansing Before Cesarean Delivery: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Sep;130(3):527-538. doi: 10.1097/AOG.0000000000002167. PMID 28796683
- [Result] Skeith AE, Niu B, Valent AM, Tuuli MG, Caughey AB. Adding Azithromycin to Cephalosporin for Cesarean Delivery Infection Prophylaxis: A Cost-Effectiveness Analysis. Obstet Gynecol. 2017 Dec;130(6):1279-1284. doi: 10.1097/AOG.0000000000002333. PMID 29112658
- [Result] American College of Obstetricians and Gynecologists Women's Health Care Physicians; Committee on Gynecologic Practice. Committee Opinion No. 571: Solutions for surgical preparation of the vagina. Obstet Gynecol. 2013 Sep;122(3):718-20. doi: 10.1097/01.AOG.0000433982.36184.95. PMID 23963423
- [Result] Reid VC, Hartmann KE, MCMahon M, Fry EP. Vaginal preparation with povidone iodine and postcesarean infectious morbidity: a randomized controlled trial. Obstet Gynecol. 2001 Jan;97(1):147-52. doi: 10.1016/s0029-7844(00)01087-5. PMID 11152924
- [Result] Dalton E, Castillo E. Post partum infections: A review for the non-OBGYN. Obstet Med. 2014 Sep;7(3):98-102. doi: 10.1177/1753495X14522784. Epub 2014 Feb 27. PMID 27512432
- [Result] Zuarez-Easton S, Zafran N, Garmi G, Salim R. Postcesarean wound infection: prevalence, impact, prevention, and management challenges. Int J Womens Health. 2017 Feb 17;9:81-88. doi: 10.2147/IJWH.S98876. eCollection 2017. PMID 28255256
- [Result] Haas DM, Morgan S, Contreras K, Enders S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2018 Jul 17;7(7):CD007892. doi: 10.1002/14651858.CD007892.pub6. PMID 30016540
- [Result] Kawakita T, Iqbal SN, Desale S, Fries M. Decrease in surgical site infection after cesarean delivery by implementing surgical bundle. Am J Obstet Gynecol 2018; 218:S323-S323.
- [Result] Guzman MA, Prien SD, Blann DW. Post-cesarean related infection and vaginal preparation with povidone-iodine revisited. Prim Care Update Ob Gyns 2002; 9:206-209.